CLINICAL TRIAL: NCT01512797
Title: A Randomized, Double-blind, Parallel-group, Placebo-controlled Study to Assess Efficacy, Safety and Tolerability of Sitagliptin Phosphate 100 mg as Treatment for Recurrent, Persistent or Newly Diagnosed Type 2 Diabetes After Gastric Bypass
Brief Title: Treatment of Diabetes After Gastric Bypass With Sitagliptin
Acronym: LAF33
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Blandine Laferrere (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Blandine Laferrere, Associate Professor of Medicine, Columbia University, Columbia University
Organization: Columbia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAO1107; 0000048421 (Other Grant/Funding Number: Merck & Co., Inc)
Record Dates: First submitted 2012-01-13; First posted 2012-01-19 (Estimated); Results first posted 2018-02-23 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Januvia; Sitagliptin; Diabetes; Gastric-Bypass
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (2):
- Sitagliptin phosphate (Active Comparator): 100 mg/day sitagliptin phosphate (Januvia) PO once a day for 4-5 weeks
  Interventions: Drug: Sitagliptin phosphate
- Placebo (Placebo Comparator): 1 Placebo pill / day PO once a day for 4-5 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sitagliptin phosphate — 100 mg/day orally
  Other Names: Januvia
  Arms: Sitagliptin phosphate
Other: Placebo — 1 Placebo Pill per day
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess whether Januvia (sitagliptin phosphate 100mg) is safe and effective for the treatment of Type 2 Diabetes in patients who have had Gastric Bypass.

DETAILED DESCRIPTION:
Januvia (sitagliptin phosphate 100mg) is an FDA approved medication for the treatment of Type 2 Diabetes. Sitagliptin works by inhibiting the Dipeptidyl peptidase-4 enzyme, resulting in increased active glucagon-like peptide-1 (GLP-1) levels. GLP-1 is an incretin which increases post-prandial insulin secretion. Because Gastric Bypass has also been shown to increase GLP-1 levels, this study seeks to determine the additional effect of DDP-4 inhibition on glucose control in patients who have elevated incretin levels post Gastric Bypass. The study will also assess if Januvia (Sitagliptin phosphate) is safe and well tolerated in patients after Gastric Bypass.

Recruitment and data collection for this study was started at St. Luke's Hospital in New York, NY and later moved to Columbia University Medical Center in New York, NY.

ELIGIBILITY:
Inclusion Criteria:

* Must be a resident of the NYC metropolitan area or be able to come for emergency unscheduled and regular weekly meetings in Manhattan.
* HbA1c ≥ 6.5% and ≤ 8.5 % or a fasting glucose ≥ 126 mg/dL or a random glucose ≥ 200 mg/dL at least 12 months after GBP surgery confirmed by central laboratory.
* Subject is capable and willing to give informed consent.
* Subject is otherwise in good general health, based on medical history and physical examination.
* Subject is a non smoker for at least 6 months prior to study start
* Female subjects of child bearing potential must use oral, injected or implanted hormonal methods of contraception from at least the commencement of their last normal period prior to the first administration of the challenge agent. Subjects using hormonal contraception should use a barrier method in addition from the first administration of challenge agent until their next normal period following the end of the study.

Exclusion Criteria:

* History of type 1 diabetes
* Female subject is pregnant or breastfeeding.
* Recent (< 30 days) or simultaneous participation in another clinical trial.
* Any situation that can compromise the study, including serious illness or a predictable lack of cooperation from the subject.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Blandine Laferrere, MD, Principal Investigator — New York Obesity Nutrition Research Center
Locations (1):
- New York Obesity Nutrition Research Center, Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: New York Obesity Nutrition Research Center — http://www.nyorc.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this study took place from July 2012-July 2016. Recruitment and data collection for this study was started at St. Luke's Hospital in New York, NY and later moved to Columbia University Medical Center in New York, NY.
Pre-assignment Details: 37 participants were enrolled, however only 32 participated in study procedures and demographic information collection.
Period: Overall Study
Arm/Group | Sitagliptin Phosphate | Placebo
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin Phosphate | Placebo | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (9.0) | 58.4 (7.0) | 56.3 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 4 | 4 | 8
  Hispanic White | 5 | 5 | 10
  Hispanic Black | 2 | 3 | 5
  African-American | 5 | 4 | 9
BMI [Mean (Standard Deviation); unit: kg/m2] | 32.70 (5.22) | 36.12 (7.69) | 34.41 (6.69)
HbA1c [Mean (Standard Deviation); unit: %] | 7.46 (0.78) | 6.96 (0.70) | 7.21 (0.77)
Time since Roux-en-Y gastric bypass surgery [Mean (Standard Deviation); unit: years] | 5.56 (3.77) | 5.57 (2.80) | 5.56 (3.27)
Type 2 Diabetes Mellitus duration prior to Roux-en-Y gastric bypass surgery [Mean (Standard Deviation); unit: years] | 12.9 (11.0) | 12.9 (9.3) | 12.9 (10.0)
Type 2 Diabetes Mellitus remission duration prior to study [Mean (Standard Deviation); unit: years] | 2.72 (3.10) | 2.16 (2.74) | 2.44 (2.89)
Maximum Weight before Roux-en-Y gastric bypass surgery [Mean (Standard Deviation); unit: kg] | 122.45 (19.0) | 132.89 (24.23) | 127.7 (22.1)
Weight at Roux-en-Y gastric bypass [Mean (Standard Deviation); unit: kg] | 117.5 (20.4) | 130.23 (24.6) | 123.9 (23.1)
Nadir weight after Roux-en-Y gastric bypass [Mean (Standard Deviation); unit: kg] | 73.51 (17.52) | 82.93 (13.38) | 78.22 (16.06)
Current Weight [Mean (Standard Deviation); unit: kg] | 85.98 (15.21) | 95.82 (19.71) | 90.90 (18.02)
Current weight loss since Roux-en-Y gastric bypass [Mean (Standard Deviation); unit: kg] | 31.53 (11.90) | 34.47 (13.91) | 33.00 (12.82)
Weight regain from nadir weight [Mean (Standard Deviation); unit: kg] | 12.73 (10.70) | 12.96 (10.94) | 12.84 (10.64)
Number of oral type 2 diabetes mellitus medications prior to Roux-en-Y gastric bypass [Mean (Standard Deviation); unit: number of medications] | 1.88 (0.89) | 1.75 (0.93) | 1.81 (0.90)
Participants on insulin prior to RYGB [Count of Participants; unit: Participants] | 10 | 10 | 20
Participants on insulin at time of study [Count of Participants; unit: Participants] | 3 | 4 | 7
Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 172.0 (41.5) | 151.78 (32.67) | 161.1 (37.67)
Triglycerides [Mean (Standard Deviation); unit: mg/dL] | 147.3 (123.9) | 124.7 (50.2) | 135.1 (90.6)
High-density lipoprotein [Mean (Standard Deviation); unit: mg/dL] | 54.83 (15.21) | 59.21 (29.39) | 57.19 (23.58)
Low-density lipoprotein [Mean (Standard Deviation); unit: mg/dL] | 89.18 (39.92) | 76.79 (28.24) | 82.24 (33.70)
Systolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 124.8 (21.23) | 119.1 (14.4) | 122.23 (18.4)
Diastolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 74.69 (12.26) | 69.77 (11.05) | 72.48 (11.79)

OUTCOME MEASURES:

1. Primary Outcome: Change in Postprandial Glucose Levels After Mixed Meal Test
Description: Glucose levels were measured in study participants while fasting and periodically over 3 hours after drinking a 200 kcal mixed meal test, before and after intervention (Sitagliptin or Placebo).
Time Frame: Baseline and ~4 weeks
Population: All patients completed study in both arms.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Sitagliptin Phosphate | Placebo
Number analyzed (Participants) | 16 | 16
mmol/L
  Pre-Intervention Fasting Glucose | 7.10 (1.74) | 6.52 (1.21)
  Post-Intervention Fasting Glucose | 6.44 (1.25) | 6.39 (1.23)
  Pre-Intervention 120 minute glucose | 7.51 (1.91) | 7.01 (1.38)
  Post-Intervention 120 minute glucose | 6.79 (1.65) | 6.97 (1.47)
  Pre-Intervention Average Glucose during MMT | 8.55 (1.95) | 8.12 (1.14)
  Post-Intervention Average Glucose during MMT | 7.84 (1.47) | 7.86 (1.04)
Statistical Analysis 1: Comparison: Sitagliptin Phosphate vs Placebo; Power analysis. Based on the effect of DPP-4 inhibitors in non-operated subjects with type 2 diabetes, showing a significant decrease in 120' post-prandial glucose by 1.67 mmol/L ± 0.98 mmol/L after a MMT, we estimated that a sample size of 16 subjects per group will show post-prandial glucose differences between placebo and sitagliptin group with α = 0.05 for a power > 90%; Test type: Other; p = 0.028, t-test, 2 sided — P-value refers to paired t-test comparing pre-intervention and post-intervention timepoints in Sitagliptin group

2. Primary Outcome: Change in Area Under the Curve (AUC) Glucose Levels After Mixed Meal Test
Description: Glucose levels were measured in study participants while fasting and periodically over 3 hours after drinking a 200 kcal mixed meal test, before and after intervention (Sitagliptin or Placebo). AUC was measured by trapezoidal method.
Time Frame: Baseline and ~4 weeks
Measure: Mean (Standard Deviation); unit: mmol/L/min
Arm/Group | Sitagliptin Phosphate | Placebo
Number analyzed (Participants) | 16 | 16
mmol/L/min
  Pre-Intervention Glucose AUC | 8.31 (1.92) | 7.96 (1.20)
  Post-Intervention Glucose AUC | 7.67 (1.59) | 7.75 (1.16)

3. Secondary Outcome: Effect of Sitagliptin vs Placebo on Satiety in Patients With Type 2 Diabetes After Gastric Bypass Surgery
Description: Satiety levels were measured in study participants while they were fasting and periodically over a three hour period after drinking a 200 kcal meal drink, before and after intervention via a Visual Analog Scale. Participants were asked to mark on a 0 to 150 millimeter scale their response to the following question: "How full do you feel right now?" with lower scores indicating "not full at all" and higher scores indicating "extremely full."
Time Frame: Baseline and ~4 weeks
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Sitagliptin Phosphate | Placebo
Number analyzed (Participants) | 16 | 16
mm
  Pre-Intervention fasting satiety level | 51.94 (87.40) | 49.06 (39.36)
  Post-Intervention fasting satiety level | 22.38 (22.03) | 58.50 (113.23)
  Pre-Intervention 180 minute glucose | 37.81 (40.95) | 50.50 (59.37)
  Post-Intervention 180 minute glucose | 43.69 (43.85) | 103.75 (198.35)

4. Secondary Outcome: Occurrence of Side Effects In Relation to Sitagliptin
Description: Side effects to Sitagliptin or Placebo were measured in study participants via Sigstad score questionnaire, while fasting and periodically during a 3 hour period after drinking a 200 kcal meal drink, before and after intervention. The Sigstad scoring system is based on the participants report of the occurrence of 16 symptoms suggestive of the dumping syndrome. Each symptom is given a different score. For example, desire to sit down (+4), breathlessness (+3), dizziness (+2), nausea (+1), vomiting (-4) etc.The scale can range from -5 to 34. Scores greater than or equal to 7, after glucose intake, are considered diagnostic of dumping syndrome.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on Sigstad scale
Arm/Group | Sitagliptin Phosphate | Placebo
Number analyzed (Participants) | 16 | 16
units on Sigstad scale
  Pre-Intervention Average Sigstad Score | 2.15 (1.97) | 5.58 (3.41)
  Post-Intervention Average Sigstad Score | 2.24 (2.34) | 4.40 (3.10)

5. Secondary Outcome: Active GLP-1
Description: Active GLP-1 (Fasting and during a Mixed Meal Test). The Change in Fasting Active GLP-1 refers to the change in fasting active GLP-1 from pre-intervention time point to post-intervention time point. The Change in Peak Active GLP-1 refers to the change in the peak active GLP-1 level from the pre-intervention time point to post-intervention time point.
Time Frame: Pre-Intervention and Post-Intervention
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Sitagliptin Phosphate | Placebo
Number analyzed (Participants) | 16 | 16
pmol/L
  Change in Fasting Active GLP-1 | 1.45 (2.59) | -0.22 (0.88)
  Change in Peak Active GLP-1 | 22.08 (15.46) | 2.97 (10.44)

ADVERSE EVENTS:
Time Frame: Over 6 weeks (the time period a participant was involved in the study).
Arm/Group | Sitagliptin Phosphate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

LIMITATIONS AND CAVEATS:
Study of short duration, designed as proof of concept. Absorption of sitagliptin may have been variable amongst subjects. The groups were small and the data cannot be extrapolated to a larger group of individuals with wide range of diabetes control.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No